CLINICAL TRIAL: NCT01329458
Title: Contrast Enhanced Ultrasound for the Evaluation of Focal Liver Lesions - a Multi-center Study on the Usefulness in the Clinical Practice
Brief Title: Contrast Enhanced Ultrasound For The Evaluation Of Focal Liver Lesions
Acronym: HepFocUS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Societatea Romana de Ultrasonografie in Medicina si Biologie (Other)
Collaborators: Centrul de Cercetare in Gastroenterologie si Hepatologie, Craiova (Unknown); Clinica de Gastroenterologie si Hepatologie, UMF Timisoara (Unknown); Institutul Regional de Gastroenterologie & Hepatologie Prof. dr. Octavian Fodor (Other); Institutul Clinic Fundeni (Other); Clinica de Gastroenterologie Constanta (Unknown)
Responsible Party: Socaciu Mihai, Societatea Romana de Ultrasonogragrafie in Medicina si Biologie
Other Study IDs: HepFocUS
Record Dates: First submitted 2011-04-02; First posted 2011-04-06 (Estimated); Last update posted 2011-04-06 (Estimated); Status verified 2011-04

CONDITIONS: Focal Nodular Hyperplasia of Liver; Toxic Liver Disease With Focal Nodular Hyperplasia; Liver Metastases
Keywords: FLL; CEUS; SonoVue; HCC; Liver metastases; Hemangiomas; FNH
MeSH Terms: conditions — Hemangioma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Focal liver lesions: Focal liver lesions: patients discovered with new, uncharacteristic focal liver lesions at standard ultrasound

SUMMARY:
The aim of the study is to assess the value of contrast enhanced ultrasound in the evaluation of de novo focal liver lesions in clinical practice, in a prospective multi-center design.

DETAILED DESCRIPTION:
Focal liver lesions (FLL) are quite frequently discovered in daily practice at routine ultrasound and sometimes require the use of extensive investigations for a correct diagnosis, thus increasing the costs and duration of diagnosis. On the other hand, due to screening strategies for patients with liver cirrhosis, FLL are discovered very early in these patients, and they must be evaluated in order to establish a therapeutic strategy (including transplantation, surgical resection or percutaneous echoguided procedures).

Contrast enhanced ultrasound (CEUS) using second generation contrast agents is a relatively new imaging modality that allows the characterization of FLL and allows a positive diagnosis based on the vascular pattern of the lesion. The advantages of this method are the low cost as compared with other imaging modalities and the fact that it can be performed immediately after standard abdominal ultrasound, so approximately 5 minutes after CEUS (the total duration of this investigation) a confident diagnosis can be obtained.

The place of CEUS in the diagnostic algorithm of FLL is not very well established. The European Federation of Societies for Ultrasound in Medicine and Biology (EFSUMB) issued the first Guidelines regarding the use of CEUS in 2004, revised in 2008, in which the main indications of this method are presented.

The purpose of this study is to establish the value of CEUS in the evaluation of de novo FLL in clinical practice.

The study will include patients discovered with de novo FLL at standard ultrasound in which the ultrasound study is not conclusive for the positive diagnosis (the patients with simple cysts or known FLL under CEUS follow up will be excluded form the study). The standard ultrasound will be followed by the contrast study using SonoVue® (Bracco, Italy) as contrast agent. The amount of contrast agent will be documented in every patient (it depends on the ultrasound machine used and the suspected diagnosis). The examination will be performed using the dedicated contrast software of each ultrasound machine used in the study. The investigators shall also document in every patient: the indication for CEUS study, a short history including the presence of chronic hepatopathies or malignancies, the ultrasound machine used and the operator. Each examination will last about 5 min after bolus injection and will be documented by 4 video files no longer than 30 seconds each, containing: The standard study, the arterial phase, the portal phase and the late phase. Additional loops can be stored whenever it is considered necessary.

A CEUS diagnosis will be established based on the contrast study. This will be compared with the final diagnosis which will be established based on all available imaging and clinical data: computer tomography, MRI, biopsy, follow up information. A CEUS examination will be considered conclusive if, following contrast, the FLL had a typical enhancement pattern according to the EFSUMB guidelines, and inconclusive if the enhancement pattern of the lesions was not in concordance with this guide.

The stored loops will be also revised by different operators. The study design is prospective, multi-center and will be approved by the ethical review board.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with de novo FLL at standard ultrasound
* age > 18 years, male and female gender
* informed consent for the contrast enhanced study

Exclusion Criteria:

* patients with contraindication for contrast enhanced study: subjects with acute cardiac infarction, with class III/IV cardiac insufficiency, with rhythm disorders and pregnant women
* Patients diagnosed with simple cysts at standard ultrasound (biliary of hydatid)
* Patients with known FLL, for example after percutaneous treatment, in which the contrast study is used for the follow up of the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients included in the study will be patients discovered with FLL at standard ultrasound. The focal lesions will be characterized by CEUS and the diagnosis established will be compared with the final diagnosis of the patient.
  The final diagnosis will be established based on all available imaging and clinical data: computer tomography, MRI, biopsy, follow up information.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2010-12; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
evaluation of contrast enhanced ultrasound in the assessment of de novo focal liver lesions | 12 months evaluation
  A CEUS examination will be considered conclusive if, following contrast, the FLL had a typical enhancement pattern according to the EFSUMB guidelines, and inconclusive if the enhancement pattern of the lesions was not in concordance with this guide.

CONTACTS AND LOCATIONS:
Locations (5):
- Romania (5):
  - Institutul Clinic Fundeni, Bucharest
  - Institutul Regional de Gastroenterologie-Hepatologie "Octavian Fodor",, Cluj-Napoca
  - Clinica de Gastroenterologie Constanta, Constanța
  - Centrul de Cercetare in Gastroenterologie si Hepatologie, Craiova
  - Clinica de Gastroenterologie si Hepatologie, Timișoara

REFERENCES:
- [Background] Albrecht T, Blomley M, Bolondi L, Claudon M, Correas JM, Cosgrove D, Greiner L, Jager K, Jong ND, Leen E, Lencioni R, Lindsell D, Martegani A, Solbiati L, Thorelius L, Tranquart F, Weskott HP, Whittingham T; EFSUMB Study Group. Guidelines for the use of contrast agents in ultrasound. January 2004. Ultraschall Med. 2004 Aug;25(4):249-56. doi: 10.1055/s-2004-813245. No abstract available. PMID 15300497
- [Background] Claudon M, Cosgrove D, Albrecht T, Bolondi L, Bosio M, Calliada F, Correas JM, Darge K, Dietrich C, D'Onofrio M, Evans DH, Filice C, Greiner L, Jager K, Jong Nd, Leen E, Lencioni R, Lindsell D, Martegani A, Meairs S, Nolsoe C, Piscaglia F, Ricci P, Seidel G, Skjoldbye B, Solbiati L, Thorelius L, Tranquart F, Weskott HP, Whittingham T. Guidelines and good clinical practice recommendations for contrast enhanced ultrasound (CEUS) - update 2008. Ultraschall Med. 2008 Feb;29(1):28-44. doi: 10.1055/s-2007-963785. No abstract available. PMID 18270887
- [Background] Strobel D, Seitz K, Blank W, Schuler A, Dietrich C, von Herbay A, Friedrich-Rust M, Kunze G, Becker D, Will U, Kratzer W, Albert FW, Pachmann C, Dirks K, Strunk H, Greis C, Bernatik T. Contrast-enhanced ultrasound for the characterization of focal liver lesions--diagnostic accuracy in clinical practice (DEGUM multicenter trial). Ultraschall Med. 2008 Oct;29(5):499-505. doi: 10.1055/s-2008-1027806. PMID 19241506
- [Background] Tranquart F, Correas JM, Ladam Marcus V, Manzoni P, Vilgrain V, Aube C, Elmaleh A, Chami L, Claudon M, Cuilleron M, Diris B, Garibaldi F, Lucidarme O, Marion D, Beziat C, Rode A, Tasu JP, Trillaud H, Bleuzen A, Le Gouge A, Giraudeau B, Rusch E. [Real-time contrast-enhanced ultrasound in the evaluation of focal liver lesions: diagnostic efficacy and economical issues from a French multicentric study]. J Radiol. 2009 Jan;90(1 Pt 2):109-22. doi: 10.1016/s0221-0363(09)70089-7. French. PMID 19212279
- [Background] Braun B. Focal liver processes: "better is the enemy of good": CEUS in the fast lane. Ultraschall Med. 2009 Aug;30(4):329-32. doi: 10.1055/s-0028-1109693. Epub 2009 Aug 17. No abstract available. English, German. PMID 19688667
- [Background] Wilson SR, Greenbaum LD, Goldberg BB. Contrast-enhanced ultrasound: what is the evidence and what are the obstacles? AJR Am J Roentgenol. 2009 Jul;193(1):55-60. doi: 10.2214/AJR.09.2553. PMID 19542395
- [Background] Trillaud H, Bruel JM, Valette PJ, Vilgrain V, Schmutz G, Oyen R, Jakubowski W, Danes J, Valek V, Greis C. Characterization of focal liver lesions with SonoVue-enhanced sonography: international multicenter-study in comparison to CT and MRI. World J Gastroenterol. 2009 Aug 14;15(30):3748-56. doi: 10.3748/wjg.15.3748. PMID 19673015
- [Background] Quaia E, Calliada F, Bertolotto M, Rossi S, Garioni L, Rosa L, Pozzi-Mucelli R. Characterization of focal liver lesions with contrast-specific US modes and a sulfur hexafluoride-filled microbubble contrast agent: diagnostic performance and confidence. Radiology. 2004 Aug;232(2):420-30. doi: 10.1148/radiol.2322031401. PMID 15286314
- [Background] von Herbay A, Vogt C, Willers R, Haussinger D. Real-time imaging with the sonographic contrast agent SonoVue: differentiation between benign and malignant hepatic lesions. J Ultrasound Med. 2004 Dec;23(12):1557-68. doi: 10.7863/jum.2004.23.12.1557. PMID 15557299
- [Derived] Sirli R, Sporea I, Popescu A, Danila M, Sandulescu DL, Saftoiu A, Moga T, Sparchez Z, Cijevschi C, Mihai C, Ioanitescu S, Nedelcu D, Iacob N, Miclaus G, Brisc C, Badea R. Contrast-enhanced ultrasound for the assessment of focal nodular hyperplasia - results of a multicentre study. Med Ultrason. 2021 May 20;23(2):140-146. doi: 10.11152/mu-2912. Epub 2021 Apr 22. PMID 33945596
- [Derived] Sporea I, Sandulescu DL, Sirli R, Popescu A, Danila M, Sparchez Z, Mihai C, Ioanitescu S, Moga T, Timar B, Brisc C, Nedelcu D, Saftoiu A, Enachescu V, Badea R. Contrast-Enhanced Ultrasound for the Characterization of Malignant versus Benign Focal Liver Lesions in a Prospective Multicenter Experience - The SRUMB Study. J Gastrointestin Liver Dis. 2019 Jun 1;28:191-196. doi: 10.15403/jgld-180. PMID 31204417
- [Derived] Sirli R, Sporea I, Sandulescu DL, Popescu A, Danila M, Saftoiu A, Sparchez Z, Badea R. Contrast enhanced ultrasound for the diagnosis of liver hemangiomas - results of a Romanian multicentre study. Med Ultrason. 2015 Dec;17(4):444-50. doi: 10.11152/mu.2013.2066.174.csu. PMID 26649337
- See also: Related Info — http://study.umfcv.ro